CLINICAL TRIAL: NCT01712828
Title: A Phase 1, Open-Label, Two-Part, Fixed-Sequence Crossover Study to Evaluate the Effect of P-glycoprotein Inhibition on Lenalidomide Pharmacokinetics in Healthy Male Subjects
Brief Title: Effect of P-glycoprotein Inhibition on Lenalidomide Pharmacokinetics in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CC-5013-CP-011
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Lenalidomide,; Revlimid,; pharmacokinetics,; healthy male subjects
MeSH Terms: interventions — Lenalidomide; Quinidine; temsirolimus; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenalidomide plus Quinidine (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Quinidine
- Lenalidomide plusTemsirolimus and Diphenhydramine (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Temsirolimus; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Lenalidomide — 25 mg Lenalidomide capsule will be administered orally once in the first period, and once with Quinidine in the second period
Drug: Quinidine — 300 mg of Quinidine will be administered orally every 12 hours for 1 day followed by 600 mg of Quinidine administered orally every 12 hours for the next 4 consecutive days
  Arms: Lenalidomide plus Quinidine
Drug: Temsirolimus — 25 mg/mL injection of Temsirolimus will be given directly into the vein over 30 minutes once in the second period and once with Lenalidomide in the third period.
  Arms: Lenalidomide plusTemsirolimus and Diphenhydramine
Drug: Diphenhydramine — Just before Temsirolimus is given, 25 mg of Diphenhydramine (Benadryl) will be given directly into the vein to decrease chances of an allergic reaction to Temsirolimus.
  Other Names: Benadryl
  Arms: Lenalidomide plusTemsirolimus and Diphenhydramine

SUMMARY:
To find out if the blood level of lenalidomide can be changed when a drug that prevents p-glycoprotein (a protein naturally present in the body that helps carry substances across cell membranes that is found in many parts of the body like the intestines, liver, and kidneys) from working (called a P-gp inhibitor) when taken together with lenalidomide. The study is also trying to find out if blood level of temsirolimus can be changed when a subject takes lenalidomide together with temsirolimus.

DETAILED DESCRIPTION:
This will be a single-center, open label, 2-part study. Part 1 will be a two-period, fixed-sequence crossover study with lenalidomide alone in Period 1, followed by lenalidomide in combination with quinidine in Period 2. Part 2 will be a fixed-sequence, three-period, crossover study with lenalidomide alone in Period 1, temsirolimus (via direct intravenous infusion) in Period 2, and lenalidomide in combination with temsirolimus (via direct intravenous infusion) in Period 3. Diphenhydramine (given via intravenous injection) will be administered shortly before temsirolimus in order to decrease the chances of an allergic reaction to temsirolimus. Part 1 and Part 2 will be conducted at the same time. Subjects can only participate in either Part 1 or Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign a written informed consent form prior to any study-related procedures being performed.
* Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
* Healthy male volunteer of any race between 18 to 65 years of age (inclusive), and in good health as determined by a physical exam.
* Agree to use barrier contraception (i.e., condoms not made of natural (animal) membrane [e.g., latex or polyurethane condoms are acceptable]) when engaging in sexual activity with a female of child-bearing potential while on study drug, and for at least 90 days after the last dose of study drug.
* Must have a body mass index between 18 and 33 kg/m2 (inclusive).
* Clinical laboratory tests must be within normal limits or acceptable to the principal investigator.
* Must have confirmation of normal renal function (defined as an estimate glomerular filtration rate >90 mL/min).
* Must be afebrile, with supine systolic blood pressure: 90 to 140 mmHg, supine diastolic blood pressure: 60 to 90 mmHg, and pulse rate: 40 to 110 bpm.
* Must have a normal or clinically acceptable 12-lead electrocardiogram, with a QTcF (Fridericia's correction formula) value ≤ 430 msec.
* Must refrain from sperm donations for the entire duration of the study, and for at least 90 days after the last dose of study drug.

Exclusion Criteria:

* History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, known hypersensitivity to a member of the class of immunomodulatory drugs (IMiDs®), temosirolimus, sirolimus, polysorbate 80, diphenhydramine, or to any other component (or excipients) of Torisel®, or other major disorders.
* Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
* Used any prescribed systemic or topical medication within 30 days of the first dose administration, unless Sponsor agreement is obtained.
* Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless Sponsor agreement is obtained.
* Used any prescribed, or non-prescribed, systemic or topical medication that is a CYP3A inhibitor or inducer within 30 days of first dose administration. (refer to (http://medicine.iupui.edu/clinpharm/ddis/p450_Table_Oct_11_2009.pdf)
* Has any surgical or medical conditions (excluding appendectomy) possibly affecting drug absorption, distribution, metabolism and excretion, e.g., bariatric procedure.
* Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
* History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.
* History of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dosing, or positive alcohol screen.
* Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb), or have a positive result to the test for HIV antibodies at Screening.
* Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
* For Part 2 only: has total bilirubin ≥ 1.5x upper limit of normal

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Lenalidomide PK-AUC (0-24) | Up to 21 days
  Area under the plasma concentration-time curve from time zero to 24 hours post dose
Lenalidomide PK-(Cmax) | Up to 21 days (including washout phase)
  Maximum observed plasma concentration
Lenalidomide PK-(Tmax) | Up to 21 days
  Time to maximum observed plasma concentration
Lenalidomide PK-AUC(0-t) | Up to 21 days
  Area under the plasma concentration-time curve from time zero to time t, where t is the last measurable time point
Lenalidomide PK-AUC(0-∞) | Up to 21 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Lenalidomide PK-(T1/2) | Up to 21 days
  Estimate of the terminal elimination half-life in plasma
Temsirolimus and Sirolimus PK-AUC (0-24) | Up to 38 days
  Area under the plasma concentration-time curve from time zero to 24 hours post dose
Temsirolimus and Sirolimus PK-(Cmax) | Up to 38 days
  Maximum observed plasma concentration
Temsirolimus and Sirolimus PK-(Tmax) | Up to 38 days
  Time to maximum observed plasma concentration
Temsirolimus and Sirolimus PK-(AUC 0-t) | Up to 38 days
  Area under the plasma concentration-time curve from time zero to time t, where t is the last measurable time point

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 6 weeks
  Safety monitoring will be done by regular adverse event assessment, concomitant medication, clinical laboratory tests, physical exams, ECGs, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation
Locations (1):
- Covance Clinical Research Unit Dallas, Dallas, Texas, United States

REFERENCES:
- See also: Related Info — http://us.testwiththebest.com/find-our--clinics/our-dallas-clinic.html